CLINICAL TRIAL: NCT05083143
Title: The Impact of the COVID-19 Pandemic on Oncologic Outcomes of Testicular Cancer
Brief Title: The Impact of the COVID-19 Pandemic on Testicular Cancer
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: COVIDTC2021
Record Dates: First submitted 2021-10-17; First posted 2021-10-19 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Testicular Cancer; COVID-19
Keywords: Testicular Cancer; COVID-19; Radical Orchiectomy
MeSH Terms: conditions — Testicular Neoplasms; COVID-19 | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Testicular Cancer: Patients diagnosed with testicular cancer in the COVID-19 period
  Interventions: Behavioral: COVID-19 pandemic
- PreCOVID-19 Testicular Cancer: Patients diagnosed with testicular cancer before the COVID-19 period
  Interventions: Behavioral: COVID-19 pandemic

INTERVENTIONS:
Behavioral: COVID-19 pandemic — Patients diagnosed with testicular cancer in the urology clinic during and before the COVID-19 pandemic will be retrospectively evaluated and compared.

SUMMARY:
In this study, investigators aim to reveal how the COVID-19 pandemic process affects testicular cancer presentations, tumor stages, the time elapsed between diagnosis and intervention, tumor recurrence and progression, which are oncological outcomes.

DETAILED DESCRIPTION:
The rapid spread of the 2019 coronavirus disease (COVID-19) caused by a novel betacoronavirus known as the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) has had dramatic effects on individuals and health systems around the world. Beyond those infected with SARS-CoV-2,the intense demand for limited health system resources has led to reduced capacity, rapid depletion of healthcare systems and hospitals becoming a source of virus transmission.

Urology associations and reference centers have issued recommendations to inform urology care during the COVID-19 outbreak. It is essential that urologists give priority to patient safety. Potential delays in the diagnosis and treatment of urological conditions and the additional burden on healthcare resources must be balanced against the risks of exposure to COVID-19. While this situation aims to conserve healthcare resources, it has created the risk of delaying cancer treatment. As a result, the transformation of health services and the increasing interest of the public in avoiding exposure to the disease has led to a decrease in the number of hospital admissions.

The effects of the pandemic on patients with testicular cancer due to a decrease in emergency room and urology clinic admissions are not clear. During theCOVID-19 outbreak, the EAU (European Association of Urology) panel of testicular cancer published an evidence-based guideline. According to this guideline, four priority groups were formed and a certain period of delaying treatment was defined for patients in each group according to their priorities.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with testicular cancer in the urology clinic.

Exclusion Criteria:

* Previous history of genitourinary system tumor
* Previous history of radiotherapy or chemotherapy

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with testicular cancer in the urology clinic
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Rate of tumor stages | 2 month
  Rate of tumor stages in patients who diagnosed with testicular cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yıldız, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yue H, Bai X, Wang J, Yu Q, Liu W, Pu J, Wang X, Hu J, Xu D, Li X, Kang N, Li L, Lu W, Feng T, Ding L, Li X, Qi X; Gansu Provincial Medical Treatment Expert Group of COVID-19. Clinical characteristics of coronavirus disease 2019 in Gansu province, China. Ann Palliat Med. 2020 Jul;9(4):1404-1412. doi: 10.21037/apm-20-887. Epub 2020 Jul 13. PMID 32692208
- [Background] Moul JW, Paulson DF, Dodge RK, Walther PJ. Delay in diagnosis and survival in testicular cancer: impact of effective therapy and changes during 18 years. J Urol. 1990 Mar;143(3):520-3. doi: 10.1016/s0022-5347(17)40007-3. PMID 2304163
- [Background] Wallis CJD, Novara G, Marandino L, Bex A, Kamat AM, Karnes RJ, Morgan TM, Mottet N, Gillessen S, Bossi A, Roupret M, Powles T, Necchi A, Catto JWF, Klaassen Z. Risks from Deferring Treatment for Genitourinary Cancers: A Collaborative Review to Aid Triage and Management During the COVID-19 Pandemic. Eur Urol. 2020 Jul;78(1):29-42. doi: 10.1016/j.eururo.2020.04.063. Epub 2020 May 3. PMID 32414626